CLINICAL TRIAL: NCT01523327
Title: Association of Maternal Uric Acid With Maternal Condition and Fetal Outcome in Pregnant Women With Hypertension
Brief Title: Study of Association Between Maternal Uric Acid , Maternal and Fetal Outcome in Pregnant Women With Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, nermin marzouk agaibi, Nermin Marzouk Agaibi, Ain Shams Maternity Hospital
Other Study IDs: ainshamsMH
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Uric Acid and Hypertension in Pregnancy
Keywords: Uric acid
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: 40 pregnant Women with hypertension who have uric acid level more than 6 mg per dL.
  Interventions: Other: measuring protein creatinin ratio,serum uric acid
- B: 40 pregnant women with hypertension who have uric acid level less than 6 mg per dl.
  Interventions: Other: measuring protein creatinin ratio,serum uric acid

INTERVENTIONS:
Other: measuring protein creatinin ratio,serum uric acid — A non-deproteinized Jaffe reaction is employed to measure creatinine and urinary protein measured by an automated colorimetric assay using pyrogallol red and sodium molybdate.
  Measuring of serum uric acid by(2,4,6-tribromo-3-hydroxybenzoic acid)TBHBA by uricase method.

SUMMARY:
Association of maternal uric acid with maternal condition and fetal outcome in pregnant women with hypertension.

DETAILED DESCRIPTION:
Association of maternal uric acid with maternal condition(renal function,liver function,...ect.) and fetal outcome(birth weight,APGER score) in pregnant women with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-40 years old
* Gestational age:28-42 weeks gestation singleton pregnancy of living fetus
* Non smoker

Exclusion Criteria:

* women who refuse the study
* Any medical or obstetric disorders especially D.M.,renal disease,hepatic, cardiac disorders or gout arthritis, other than hypertension if present.
* Previously elevated uric acid level.
* Hemolytic or sickle cell anemia,urinary tract infection.
* Use of diuretics or anti-inflammatory drugs.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include 80 pregnant ladies with hypertension admitted to the maternity ward of the hospital who will be divided into two groups according to their uric acid level.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Saeedeldin Elsafty, assistant lecture, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain shams maternity hospital, Cairo, Egypt

REFERENCES:
- [Result] MATSELIUKH BP. [TRANSMISSION OF CERTAIN BIOCHEMICAL PROPERTIES IN ACTINOMYCETES BY MEANS OF DNA UNDER CONDITIONS OF HETEROTRANSFORMATION]. Mikrobiol Zh. 1963;25:3-6. No abstract available. Russian. PMID 14071979
- [Result] Paula LG, da Costa BE, Poli-de-Figueiredo CE, Antonello IC. Does uric acid provide information about maternal condition and fetal outcome in pregnant women with hypertension? Hypertens Pregnancy. 2008;27(4):413-20. doi: 10.1080/10641950801955709. PMID 19003642
- See also: does+uric+acid+provide+information+about+maternal+condition+and+fetal+outcome+in+pregnant+women+with+hypertension&TransSchema=title&cmd=detailssearch — http://www.ncbi.nlm.nih.gov/pubmed?term=does+uric+acid+provide+information+about+maternal+condition+and+fetal+outcome+in+pregnant+women+with+hypertension&TransSchema=title&cmd=detailssearch
- See also: does+uric+acid+provide+information+about+maternal+condition+and+fetal+outcome+in+pregnant+women+with+hypertension&TransSchema=title&cmd=detailssearch — http://www.ncbi.nlm.nih.gov/pubmed?